CLINICAL TRIAL: NCT04217681
Title: Non-pharmacological Treatments (Self-hypnosis/Self-care and Music-therapy) for Non-malignant and Malignant Pain : a Randomized Study
Brief Title: Non-pharmacological Treatments for Non-malignant and Malignant Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/85-B
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Comparison of Treatment for Chronic Non-malignant and Malignant Pain
Keywords: chronic pain; cancer; self-hypnosis; self-care; music-therapy; motivation
MeSH Terms: conditions — Chronic Pain; Neoplasms

STUDY DESIGN:
Intervention Model Description: Each patients will have a medical consultation and will have to fill-in questionnaires (T0). After, patients will have to participate in a 5-session psycho-education programme. After, the care staff will have a multidisciplinary discussion and will randomize the participants to different treatment groups : self-hypnosis/self-care and music/self-care. Another group will be included but will not be randomized because it includes patients who demand to learn self-hypnosis/self-care (non-malignant and malignant pain). After, participants will receive a 7 months (2 hours session a month) learning program of self-hypnosis/self-care animated by a therapist specialized in hypnosis or music/self-care (identical procedure but the hypnosis is replaced by music) at the end if which they will complete the same questionnaire (T2). A follow-up at 6 (T3) and 12 (T4) months will also be conducted to account for any long term effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-hypnosis/self-care group (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care
- Music/self-care (Experimental): It is a 7-months 2 hours-session (1 session per month) of music/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. At the end of each session, patients are invited to listen to a relaxing melody of 15 minutes. This melody was composed by a professional musico-therapist. A CD with the audiotaped melody is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Music/self-care
- Self-hypnosis/self-care motivation (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care motivation
- Self-hypnosis/self-care malignant pain (Experimental): It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care malignant pain

INTERVENTIONS:
Behavioral: Self-hypnosis/self-care — It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Arms: Self-hypnosis/self-care group
Behavioral: Music/self-care — It is a 7-months 2 hours-session (1 session per month) of music/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. At the end of each session, patients are invited to listen to a relaxing melody of 15 minutes. This melody was composed by a professional musico-therapist. A CD with the audiotaped melody is given to each patient so that they can practice also every day.
  Arms: Music/self-care
Behavioral: Self-hypnosis/self-care motivation — It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Arms: Self-hypnosis/self-care motivation
Behavioral: Self-hypnosis/self-care malignant pain — It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercise is conducted at the end of each session. A CD with the audiotaped hypnosis exercise is given to each patient so that they can practice also every day.
  Arms: Self-hypnosis/self-care malignant pain

SUMMARY:
Chronic pain concerns one in four adults in Belgium. Because of the psychological and social repercussions, a biopsychosocial approach is necessary in order to improve the quality of life of people suffering from chronic pain. Non-pharmacological techniques such as hypnosis, self-care learning and music-therapy are gaining more and more interest in the scientific field. Indeed, several studies have shown a reduction in psychological distress and an improvement in global quality of life after having learned self-hypnosis/self-care. Furthermore, other studies focusing on music as a treatment for chronic pain highlight an analgesic effect of music over pain and a reduction of common comorbidities. Nevertheless, only few studies aim at comparing these techniques to each other. The aim of our study would be to compare a 7 months learning program of self-hypnosis/self-care, music-therapy/self-care, motivation to learn self-hypnosis/self-care in order to highlight the most efficient treatment for chronic pain. Furthermore, we will include another type of chronic pain i.e. cancer pain to understand if self-hypnosis/self-care's impact is different in the other type of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Fluency in French
* Chronic pain diagnosis (malignant and non-malignant)

Exclusion Criteria:

* Neurologic disorder
* Psychiatric disorder
* Drug addiction
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain description | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of slef-hypnosis/self-care on pain description will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (no pain) to 10 (worst pain).
Change in sleep | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care upon the severity of insomnia will be assessed by means of the "Insomnia Severity Index" (Morin et al., 2001). Scale ranging from 0 (none) to 4 (very severe).
Change in anxiety | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on anxiety will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in depression | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on depression will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Change in pain disability | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on pain disability will be assessed by means of the "Pain Disability Index" (PDI, Tait et al., 1990). Scale ranging from 0 (no difficulties) to 10 (a lot of difficulties).
Change in attitudes and beliefs about pain | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the attitudes and beliefs about pain will be assessed my means of the "Survey of Pain Attitudes" (SOPA, Jensen & Karoly, 1987). Scale ranging from 0 (totally wrong) to 10 (totally right).
Change in quality of life | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the quality of life will be assessed by means of the "Short Form-36"(SF-36, Ware et al., 1988). Each item is balanced to obtain a score between 0 (worst quality) to 100 (maximum quality).
Change in locus of control | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the locus of control will be assessed my means og the "Multidimensional Health Locus of Control" (MHLC, Wallston et al., 1978). Scale ranging from 1 (no agreement) to 4 (agreement).
Change of the impact of pain | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on the impact of pain in individual's life, quality of social support and general activity, will be assessed my means of the "Multidimensional Pain Index" (PDI, Kerns et al., 1985). Scale ranging from 0 (none) to 6 (a lot).
Change in generic health | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of self-hypnosis/self-care on generic health will be assessed by the "EuroQol 5 Dimensions" questionnaire (EQ-5D, Health Policy, 1990). Scale ranging from 1 (no problems) to 3 (extreme problems).
Change in health status | Day 0 (before the intervention), up to 7 months (right after the intervention), up to 13 months (6 months follow-up), up to 19 months (12 months follow-up)
  The impact of Self-hypnosis/self-care on global health status will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (worst health status) to 100 (best health status).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Liège, Liège, Belgium